CLINICAL TRIAL: NCT00805454
Title: A Phase I, Open-Label,Positron Emission Tomography (PET) Study Healthy Subjects Following a Single Oral Dose of OPC-34712
Brief Title: Positron Emission Tomagraphy (PET) Study Following a Single Oral Dose of OPC-34712
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Otsuka Pharmaceutical Development & Commercialization, Inc. (Industry)
Collaborators: Otsuka Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Patricia Bricmont, PhD, Associate Director Clinical Pharmacology, Otsuka Pharmaceutical Development & Commercialization, Inc.
Masking: None | Purpose: Basic Science
Other Study IDs: 331-07-202
Record Dates: First submitted 2008-12-04; First posted 2008-12-09 (Estimated); Last update posted 2010-05-07 (Estimated); Status verified 2010-05

CONDITIONS: Schizophrenia
Keywords: Healthy Volunteers; Phase I; Pet Scan
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: OPC-34712 — Single oral dose, 0.5 to 25 mg

SUMMARY:
Determine the degree of striatal D2 receptor occupancy induced by OPC-34712 at differenht dose levels in healthy volunteers.

DETAILED DESCRIPTION:
Subjects will receive a dose of study medication and will undergo a PET scan at 4 hrs and 23.5 hours post dose. Subjects will remain in the clinic from Day-1 to Day 7 for PK sample collection and safety monitoring. Subjects will return to the clinic on Day 10 for a follow-up safety assessment.

ELIGIBILITY:
Inclusion Criteria:

* Males and non-child bearing potential females between 18 and 45 years of age, inclusive.
* BMI between 19 and 32 kg/m2, inclusive.

Exclusion Criteria:

* Condition or history which may present a safety concern to the subject or interfere with outcome variables.
* History of or current drug or alcohol abuse, hepatitis, AIDS, or drug allergy.
* Use of prescription, over-the-counter, or herbal medication, or vitamin supplements within 14 days or antibiotics within 30 days.
* Use of tobacco products or daily exposue to second hand smoke.
* Blood pressure higher than 140/90 mmHg or lower than 100/50 mmHg: heart rate outside 40 to 90 beats/minute.
* History of serious mental disorder.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2008-12; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
Pharmacodynamic: Percent occupancy of D2 receptor, as judged by PET scan. | 10 days

SECONDARY OUTCOMES:
Measure safety: adverse events, vital signs, ECGs, and clinical laboratory tests | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Dean Wong, MD,PhD, Principal Investigator — Johns Hopkins University, Baltimore,MD 21287; Stephen Bart, MD, Principal Investigator — SNBL, Baltimore,MD 21201

REFERENCES:
- [Derived] Wong DF, Raoufinia A, Bricmont P, Brasic JR, McQuade RD, Forbes RA, Kikuchi T, Kuwabara H. An open-label, positron emission tomography study of the striatal D2/D3 receptor occupancy and pharmacokinetics of single-dose oral brexpiprazole in healthy participants. Eur J Clin Pharmacol. 2021 May;77(5):717-725. doi: 10.1007/s00228-020-03021-9. Epub 2020 Nov 16. PMID 33196868